CLINICAL TRIAL: NCT06762535
Title: fMRI（Functional Magnetic Resonance Imaging,fMRI ) Study of the Neural Mechanism of rTMS(Repetitive Transcranial Magnetic Stimulation,rTMS) Stimulation of the Left Dorsolateral Prefrontal Lobe in the Treatment of Nicotine Dependence
Brief Title: fMRI Study of the Neural Mechanism of rTMS in the Treatment of Nicotine Dependence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: nicotine dependence
Record Dates: First submitted 2023-09-04; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use Disorder; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active repetitive transcranial magnetic stimulation (Active Comparator): Intervention type:Pulse field stimulator of shenzhen yingzhi co., LTD The RTMS treatment target is scheduled for the lateral frontal lobe on the left side. The TMS stimulation frequency is 10Hz, and the stimulation intensity is 100% of the motion threshold 5s, off 10s, for 10 minutes, 2,000 pulses.
  Interventions: Device: repetitive transcranial magnetic stimulation
- Sham repetitive transcranial magnetic stimulation (Sham Comparator): Intervention type:Pulse field stimulator of shenzhen yingzhi co., LTD The RTMS treatment target is scheduled for the lateral frontal lobe on the left side.
  The TMS stimulation frequency is 10Hz, and the stimulation intensity is 100% of the motion threshold 5s, off 10s, for 10 minutes, 2,000 pulses.But there's no real pulse output,Just set the same conditions.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation
- No repetitive transcranial magnetic stimulation (No Intervention): No treatment with a transcranial magnetic stimulator

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Those receiving experimental treatment will receive 10 sessions of rTMS, stimulation protocol included 10 sessions within 14 days (once a day, 5 days/week, 2 weeks, 10 Hz frequency, pulse intensity 100% of the resting motor threshold, 50 pulses per train, inter train pause of 10 s, 40 stimulation trains, 2000 pulses/ session)
  Arms: Active repetitive transcranial magnetic stimulation
Device: Sham repetitive transcranial magnetic stimulation — Those receiving experimental treatment will receive 10 sessions of rTMS, stimulation protocol included 10 sessions within 14 days (once a day, 5 days/week, 2 weeks, 10 Hz frequency, pulse intensity 100% of the resting motor threshold, 50 pulses per train, inter train pause of 10 s, 40 stimulation trains, 2000 pulses/ session).But there's no real pulse output,Just set the same conditions.
  Arms: Sham repetitive transcranial magnetic stimulation

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of treatment and the efficacy-related neural network mechanisms by stimulating the left dorsolateral prefrontal lobe with rTMS to nicotine dependent.

The main questions it aims to answer are:

* Efficacy of left dorsolateral prefrontal rTMS in the treatment of nicotine dependent subjects.
* The relationship between therapeutic effect and the internal function of the large brain networks of ECN, DMN and SN, and the changes in the interaction between the networks.

DETAILED DESCRIPTION:
Participants will randomly divided into two groups，Relevant psychological and behavioral data and fMRI data were collected first, and then rTMS was continuously treated for 2 weeks. The above data were collected again after the treatment ended, and then the follow-up was conducted for 1 month. Psychobehavioral data were collected once a week for nicotine addicts.Finally, the collected neuroimage data were analyzed to compare the difference in efficacy between the true and false treatment groups, and to clarify the relationship between the efficacy of nicotine dependent patients after rTMS treatment and the internal functions of the large brain networks of ECN, DMN and SN as well as the interaction characteristics of the networks, so as to provide a scientific basis for the development of effective individualized treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Meets the DSM-V diagnostic criteria for addiction
* Pure nicotine dependence
* Did not receive medication
* Right-handed

Exclusion Criteria:

* Patients with organic brain lesions and a history of severe head trauma
* Compliance is poor
* Multiple drug abusers
* Current or past history of mental or neurological disorders
* There was a metallic foreign object in his body
* People with pacemakers

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Smoking Survey (FTND) | Baseline, every day during treatment (up to 10 days),1 week later, 2 week later，3 week later，4week later,5week later,6week later
  The questions were set according to the time and occasion of smoking every day, and the degree of dependence on tobacco was assessed by scores. Scores range from 0 to 10, The higher the score, the greater the degree of dependence
Foundation desire assessment | Baseline, every day during treatment (up to 10 days),End of treatment:1 week later, 2 week later，3 week later，4week later
  Foundation desire assessment will be assessed with visual analogue scale,Scores range from 0 to 10, with higher numbers representing higher base desires.
Craving rating (cue) | Baseline, every day during treatment (up to 10 days),End of treatment:1 week later, 2 week later，3 week later，4week later
  Craving rating (cue) will be assessed with visual analogue scale,Scores range from 0 to 10, with higher numbers representing higher base desires.
Smoking per day | Baseline, every day during treatment (up to 10 days),1 week later, 2 week later，3 week later，4week later,5week later,6week later
  The number of smoking per day should be filled in according to the actual situation
Desired degree of quitting | Baseline, 6week later
  Desired degree of quitting will be assessed with visual analogue scale,Scores range from 0 to 10, with higher numbers representing higher base desires.
Pre-treatment Depression Self-Rating Scale (BDI) | Baseline, 6week later
  BDI will be will be assessed with visual analogue scale,Scores range from 0 to 3,The higher the score, the greater the likelihood of depression.
Pre-treatment Anxiety Rating Scale (HAMA) | Baseline, 6week later
  HAMA will be assessed with visual analogue scale,Scores range from 0 to 4,The higher the score, the greater the likelihood of anxiety.
Change of functional connectivity between dorsolateral prefrontal cortex and whole brain | Baseline, 2 week later
  Functional connectivity based on dorsolateral prefrontal cortex will be measured with magnetic resonance imaging based on blood oxygen level dependence

CONTACTS AND LOCATIONS:
Overall Officials: Menghui Yuan, phd, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

DOCUMENTS (1):
  • Study Protocol (2024-09-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT06762535/Prot_000.pdf